CLINICAL TRIAL: NCT03902184
Title: TELLOMAK: T-cell Lymphoma Anti-KIR3DL2 Therapy. An Open Label, Multicohort, Multi-center Phase II Study Evaluating the Efficacy and Safety of IPH4102/Lacutamab Alone or in Combination With Chemotherapy in Patients With Advanced T-cell Lymphoma
Brief Title: IPH4102 Alone or in Combination With Chemotherapy in Patients With Advanced T Cell Lymphoma
Acronym: TELLOMAK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPH4102-201; 2018-003969-33 (EudraCT Number); 2023-507777-18-00 (EU CTIS Number)
Record Dates: First submitted 2019-03-14; First posted 2019-04-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Relapsed/refractory Sezary Syndrome (Experimental): IPH4102 will be administered every week for 5 weeks then every 2 weeks for 10 administrations then every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Biological: IPH4102
- Cohort 2: Stage IB-IV Mycosis Fungoides, KIR3DL2 expressing (Experimental): IPH4102 will be administered every week for 5 weeks then every 2 weeks for 10 administrations then every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Biological: IPH4102
- Cohort 3: Stage IB-IV Mycosis Fungoides,KIR3DL2 non-expressing (closed) (Experimental): IPH4102 will be administered every week for 5 weeks then every 2 weeks for 10 administrations then every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Biological: IPH4102
- Cohort All comers: Stage IB-IV Mycosis Fungoides,KIR3DL2 expressing and non-expressing (Experimental): IPH4102 will be administered every week for 5 weeks then every 2 weeks for 10 administrations then every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Biological: IPH4102

INTERVENTIONS:
Biological: IPH4102 — Patients will receive a flat dose of 750mg
  Other Names: lacutamab

SUMMARY:
This is an open label, multi-cohort, and multi-center phase II study, which evaluates the clinical activity and safety of IPH4102 in Sezary Syndrome and Mycosis fungoides as single agent.

ELIGIBILITY:
Inclusion criteria

SS patients (Cohort 1):

1. Relapsed and/or refractory stage IVA, IVB SS who have received at least two prior systemic therapies;
2. Prior treatment with mogamulizumab;
3. Patients should have blood stage B2 at screening based on central evaluation by flow cytometry;
4. Feasibility of obtaining at least one skin biopsy at screening;

   MF patients (Cohorts 2 and All comers):
5. Relapsed and/or refractory stage IB, IIA, IIB, III, IV MF;
6. Only for Cohort 2: KIR3DL2 expression in at least one expressing skin lesion based on central evaluation by IHC;
7. Patients should have received at least two prior systemic therapies;
8. Feasibility of obtaining at least one skin biopsy at screening;

   Additional inclusion criteria applicable to all cohorts:
9. Male or Female, at least 18 years of age;
10. ECOG performance status ≤2;
11. The patient must have a minimum wash-out period of 3 weeks between the last dose of prior systemic therapy and the first dose of IPH4102;
12. Patients should have recovered from all non-hematological adverse events related to prior therapy to ≤ grade 1 except for alopecia;
13. Adequate baseline laboratory data:

    Hematology:
    * Hemoglobin >9 g/dL,
    * Absolute neutrophil count (ANC) ≥1,500/µL,
    * Platelets ≥100,000/µL,

    Biochemistry:
    * Bilirubin ≤1.5 X upper limit of normal (ULN) or ≤3 X ULN for patients with Gilbert's disease,
    * Serum creatinine ≤1.5 X ULN,
    * Creatinine clearance ≥30 mL/min, calculated with the Cockcroft & Gault formula,
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5 X ULN;
14. Women of childbearing potential (WOCBP): Premenopausal females who had at least one menstrual cycle in the past 12 months and capable to become pregnant. They must have a negative serum beta-HCG pregnancy test result within seven days from start of treatment;
15. Women of childbearing potential and all men (and their female partners of childbearing potential) who are sexually active must agree to use adequate method of contraception at study entry, during treatment and for at least 9 months (270 days) following the last dose of study drug;
16. Signed informed consent form prior to any protocol-specific procedures

Exclusion Criteria:

1. Patients with evidence of large cell transformation (LCT) based on central histologic evaluation at screening;
2. Receipt of live vaccines within 4 weeks prior to treatment;
3. Central nervous system (CNS) lymphoma involvement;
4. Prior administration of IPH4102;
5. Concurrent enrollment in another clinical trial, unless it is an observational (non - interventional) clinical study or the follow-up period of an interventional study;
6. Autologous stem cell transplantation less than 3 months prior to enrollment;
7. Prior allogenic transplantation;
8. Patients who have undergone major surgery ≤ 4 weeks prior to study entry;
9. Patients with known NCI CTCAE grade 3 or higher active systemic or cutaneous viral, bacterial, or fungal infection;
10. Patients who have Hepatitis B Virus infection determined as HBsAg positive and / or Hepatitis C Virus infection determined as detection of HCV RNA in serum or plasma by a sensitive quantitative molecular method;
11. Known or tested positive for human immunodeficiency virus (HIV);
12. Patients with a history of other malignancies during the past five years apart from the disease subject of this study. The following are exempt from the five-year limit: non-melanoma skin cancer, lymphomatoid papulosis, resected thyroid cancer, biopsy-proven cervical intraepithelial neoplasia, Ductal carcinoma in situ (DCIS) or cervical carcinoma in situ
13. Pregnant or breastfeeding women;
14. Known clinically significant cardiovascular disease or condition, including:

    * Class III or IV cardiovascular disease according to the New York Heart Association (NYHA) Functional Classification;
    * Any uncontrolled arrhythmia (per the investigator's discretion);
    * Uncontrolled hypertension (per the investigator's discretion).
15. Patients with autoimmune disease on systemic immunosuppressive treatment;
16. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment and/or comply with study protocol;
17. Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the first dose until study completion, an expected average of 2 years
  Using the Olsen (2011, JCO) criteria (All cohorts)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) (All cohorts) | From first dose until study completion, an expected average of 2 years
  patients with treatment-related adverse events as assessed by CTCAE v5.0
Quality of life (QoL) (All cohorts) | Through study completion, an expected average of 2 years
  Using the Skindex29 questionnaire to assesse the effects of skin disease on quality of life in three domains: Symptoms, Emotions, and Functioning
pruritus (All cohorts) | Through study completion, an expected average of 2 years
  Using Visual Analog Scale (VAS) for prutitus assessment: From 0 = No pruritus to 10 = Pruritus as bad as it could possibly be
ORR using blinded central review (Cohort 1) | From the first dose until study completion, an expected average of 2 years
  Using the Olsen (2011, JCO) criteria
Progression free survival (PFS) (All cohorts) | From the first dose until study completion, an expected average of 2 years
Overall survival (OS) (All cohorts) | From the first dose until study completion, an expected average of 2 years
PK parameters : Maximum Plasma Concentration of IPH4102 alone (All cohorts) | From the first dose until study completion, an expected average of 2 years
  Maximum Plasma Concentration (Cmax) (W1, W5)
PK parameters :Trough Concentration of IPH4102 alone (All cohorts) | From the first dose until study completion, an expected average of 2 years
  Trough Concentration (Ctrough) every 8 or 12 weeks
Immunogenicity of IPH4102 alone (All cohorts) | From the first dose until study completion, an expected average of 2 years
  A serum sample will be collected at the specified time points for evaluation of anti-drug antibodies (ADA).
Duration of Response (DOR) | From the first dose until study completion, an expected average of 2 years

CONTACTS AND LOCATIONS:
Locations (53):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Irvine Medical Center, Orange, California
  - Stanford University, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University The Feinberg School of Medicine, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Universal Dermatology, PLLC68, Fairport, New York
  - Columbia University Department of Dermatology, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Health Care Services, Fairfax, Virginia
- Austria (2):
  - Universitätsklinik für Dermatologie Medizinische Universität Graz, Graz
  - Medizinische Universitaet Wien, Vienna
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - UZ Leuven - campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
- France (10):
  - CHU de Bordeaux Saint André, Bordeaux
  - CHRU de Tours, Hôpital Trousseau, Chambray-lès-Tours
  - CHU Henri Mondor, Créteil
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Centre Hospitalier Lyon-Sud, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHRU de Montpellier - Hopital Saint Eloi, Montpellier
  - Hôpital Saint-Louis, Paris
  - Hôpital Charles Nicolle-CHU de Rouen Clinique Dermatologie, Rouen
  - IUCT Oncopôle, Toulouse
- Germany (8):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Ruhr-University Bochum, Bochum
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitaetsmedizin Mannheim GmbH, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Universitaetsklinikum Muenster, Münster
- Italy (4):
  - Institute of Hematology "Seràgnoli", Univeristy of Bologna, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - Istituto Dermopatico dell'Immacolata (IDI-IRCCS), Roma
  - Universita di Torino, Ospedale le Molinette, Turin
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Klinika Dermatologii, Wenerologii i Alergologii ul. Smoluchowskiego 17, Gdansk
  - CET Centrum Medyczne Pratia Poznan ul. Poznanska 14, Skorzewo
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Klinika Nowotworow Ukladu Chlonnego, Warsaw
- Spain (6):
  - Hospital del Mar, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Consorci Hospital General Universitari de Valencia Servicio de Dermatología, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No